CLINICAL TRIAL: NCT02755805
Title: CO-OPerative Training For Stroke Rehabilitation: A Phase II Trial Examining Meta-Cognitive Strategy Training in Acute Stroke Rehabilitation
Brief Title: CO-OPerative Training for Stroke Rehabilitation
Acronym: CO-OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Skidmore, PhD, OTR/L, Chair and Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO09010473; K12HD055931 (NIH)
Record Dates: First submitted 2016-04-25; First posted 2016-04-29 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: CO-OP; Attention Control
Keywords: Stroke; Rehabilitation; Cognition; Intervention; Strategy training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CO-OP (Experimental): Cognitive Orientation to daily Occupational Performance (CO-OP) is a strategy training approach that trains individuals to identify problems in the performance of their daily activities, develop strategies to address these problems, and monitor their own performance in the course of their daily routines. Participants use a workbook to support their application of the strategy training.
  Interventions: Behavioral: CO-OP
- Attention Control (Placebo Comparator): The attention control intervention controls for the non-specific effects of strategy training. The therapists administer the standardized and dose-matched protocol, using scripted open-ended questions to facilitate participants' reflections on their rehabilitation activities and experiences. Participants complete a daily journal, merely reviewing their rehabilitation activities.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: CO-OP
  Other Names: Strategy Training
  Arms: CO-OP
Behavioral: Attention Control
  Other Names: Reflective Listening
  Arms: Attention Control

SUMMARY:
Cognitive impairments occur frequently after stroke, and are associated with significant long-term activities of daily living (ADL) disability and poor quality of life. This research study will undertake an innovative approach addressing cognitive impairments, by examining a new patient-centered functionally-relevant rehabilitation intervention that teaches individuals with cognitive impairments to manage their deficits to reduce ADL disability.

DETAILED DESCRIPTION:
Cognitive impairments are characterized by problems sustaining attention in distracting conditions, shifting attention between different task demands, and using working memory to consistently execute intended actions, and as a result limit the ability to execute routine ADLs. Presently there are no interventions that have demonstrated robust effectiveness in reducing disability among individuals with cognitive impairments after stroke. Recent findings suggest that individuals with cognitive impairments may experience ADL disability in part because they have difficulty engaging in, and benefiting from rehabilitation programs as they are currently delivered. In other words, individuals with cognitive impairment, due to the nature of their impairments, have difficulty learning and applying adaptive strategies as they are currently provided during traditional rehabilitation training. Therefore, interventions that train individuals with cognitive impairments a new way to learn and apply adaptive strategies may help them benefit from rehabilitation programs and reduce long-term disability. Cognitive Orientation to daily Occupation Performance (CO-OP) is a strategy training approach that trains individuals to identify problems in the performance of daily activities, develop strategies to address these problems, and monitor their own performance in the course of their daily routines. Therefore, CO-OP teaches individuals to "take charge" of their rehabilitation, and develop adaptive behaviors to "work around" cognitive impairments to meet their goals. The proposed project examines whether CO-OP facilitates reductions in ADL disability and improvements in rehabilitation engagement among individuals with cognitive impairments after acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of acute stroke
* admission to acute inpatient rehabilitation
* impairment in cognitive functions (Quick Executive Interview ≥ 3)

Exclusion Criteria:

* dementia diagnosis (as indicated in the medical record)
* severe aphasia as indicated by score ≥ 2 on the Boston Diagnostic Aphasia Examination (3rd Edition) Severity Rating Scale (BDAE-3)
* current major depressive disorder (unless treated and in partial remission), bipolar or any other psychotic disorder (Primary Care Evaluation of Mental Disorders)
* drug or alcohol abuse within 3 months (Mini-International Neuropsychiatric Interview)
* anticipated length of stay less than 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Skidmore, PhD, OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data at this time.

REFERENCES:
- [Derived] Kringle EA, Terhorst L, Butters MA, Skidmore ER. Clinical Predictors of Engagement in Inpatient Rehabilitation Among Stroke Survivors With Cognitive Deficits: An Exploratory Study. J Int Neuropsychol Soc. 2018 Jul;24(6):572-583. doi: 10.1017/S1355617718000085. Epub 2018 Mar 19. PMID 29552996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 2009 to June 2012. Participants with acute stroke were enrolled in inpatient rehabilitation at Mercy and Montefiore Hospital.
Pre-assignment Details: Excluded (n=30):
  * Insufficient cognitive impairment (n=15)
  * Mood/psychotic disorder (n=5)
  * Aphasia (n=3)
  * Recent drug/alcohol abuse (n=2)
  * Primary diagnosis not stroke (n=2)
  Withdrew prior to randomization (n=3)
  * Changed mind (n=1)
  * Family reasons (n=1)
  * Unexpected discharge (n=1)
Groups:
- CO-OP: Cognitive Orientation to daily Occupational Performance (CO-OP) is a strategy training approach that trains individuals to identify problems in the performance of their daily activities, develop strategies to address these problems, and monitor their own performance in the course of their daily routines. Participants use a workbook to support their application of the strategy training.
  CO-OP
- Attention Control: The attention control intervention controls for the non-specific effects of strategy training. The therapists administer the standardized and dose-matched protocol, using scripted open-ended questions to facilitate participants' reflections on their rehabilitation activities and experiences. Participants complete a daily journal, merely reviewing their rehabilitation activities.
  Attention Control
Period: Overall Study
Arm/Group | CO-OP | Attention Control
Started | 15 | 15
Completed | 13 | 11
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Refused assessments | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CO-OP | Attention Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.87 (16.59) | 71.80 (13.19) | 67.33 (15.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 11 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 14 | 26
  African American | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Stroke onset [Mean (Standard Deviation); unit: days] — Stroke onset is calculated from date of stroke to date of study admission.
  days | 16.80 (15.58) | 18.47 (21.29) | 17.63 (18.35)
Stroke type [Number; unit: participants]
  ischemic | 10 | 11 | 21
  hemorrhagic | 5 | 4 | 9
Hemisphere [Number; unit: participants]
  right | 10 | 10 | 20
  left | 5 | 5 | 10
Stroke severity, NIHSS (National Institutes of Health Stroke Scale) [Mean (Standard Deviation); unit: units on a scale] — The NIHSS is composed of 11 items that are summed to yield a total score. Total scores range from 0 to 42; 0=no neurological impairment, 42=severe neurological impairment.
  units on a scale | 8.87 (2.77) | 5.87 (2.72) | 7.37 (3.10)
Medical burden, CIRS (Cumulative Illness Rating Scale) [Mean (Standard Deviation); unit: units on a scale] — The Cumulative Illness Rating Scale records medical problems for 14 organ systems. The severity index is computed by averaging the impairment severity for each organ system (0=no impairment, 4=severe impairment), yielding an average severity index of 0 (no medical problems) to 4 (severe medical problems).
  units on a scale | 2.37 (.47) | 2.36 (.57) | 2.37 (0.53)
Cognitive status, EXIT (Quick Executive Interview) [Mean (Standard Deviation); unit: units on a scale] — The EXIT is composed of 14 items that are summed to yield a total score ranging from 0 to 28. A total score of 0 typically indicates no executive impairment, while a total score of 28 indicates severe executive impairment.
  units on a scale | 8.13 (3.00) | 9.31 (3.54) | 8.72 (3.28)
Communication status, BDAE (Boston Diagnositic Aphasia Examination Severity Index) [Mean (Standard Deviation); unit: units on a scale] — The Boston Diagnostic Aphasia Examination is an aphasia severity rating scale ranging from 0-5, with 0 representing no usable speech or auditory comprehension and 5 representing minimal discernible speech impairments.
  units on a scale | 4.27 (1.03) | 4.67 (.62) | 4.47 (0.86)
Functional Independence Measure [Mean (Standard Deviation); unit: units on a scale] — The Functional Independence Measure contains 18 items composed of 13 motor tasks and 5 cognitive tasks. A total scores is obtained (18-126), 18 represents complete dependence/total assistance and 126 represents complete independence with daily activities.
  units on a scale | 65.27 (10.85) | 62.60 (16.56) | 63.93 (13.82)
Inhibition, CWI (Color Word Interference) [Mean (Standard Deviation); unit: units on a scale] — The Inhibition Scale raw scores are converted to norm-referenced scaled scores adjusted for age and education. These scores are aligned with a population mean of 10, and standard deviation of 3. Higher scores indicate better executive function.
  units on a scale | 4.85 (4.10) | 4.00 (2.98) | 4.39 (3.50)
Cognitive flexibility, CWI (Color Word Interference) [Mean (Standard Deviation); unit: units on a scale] — The Cognitive Flexibility Scale raw scores are converted to norm-referenced scaled scores adjusted for age and education. These scores are aligned with a population mean of 10, and standard deviation of 3. Higher scores indicate better executive function.
  units on a scale | 3.69 (2.36) | 2.73 (2.34) | 3.18 (2.36)
Depressive symptoms, HamD (Hamilton Rating Scale for Depression) [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale is composed of 17 items that are summed to yield a total score ranging from 0 to 52. A total score of 0 typically indicates no depressive symptoms; 52 indicates severe depressive symptoms.
  units on a scale | 6.71 (4.36) | 6.75 (4.53) | 6.73 (4.35)
Apathy, AES [Mean (Standard Deviation); unit: units on a scale] — The Apathy Evaluation Scale measures motivation or interest in goal-directed activities. The scale has 18 items with a total score of 18 (absence of apathy) to 72 (severe apathy).
  units on a scale | 25.79 (7.62) | 25.18 (4.40) | 25.52 (6.29)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Independence With Activities of Daily Living (Functional Independence Measure) Between Groups Over Time
Description: Difference between groups in mean scores (computed from Functional Independence Measure total scores) over time were examined with mixed effects models.
  The Functional Independence Measure contains 18 items with a total score ranging from 18-126 is obtained (18=complete dependence/total assistance with basic self-care and mobility activities; 126=complete independence with basic self-care and mobility activities). Total scores were calculated at baseline, rehabilitation discharge, month 3, and month 6 for each participant, and mean total scores were calculated fro each group at each time point.
Time Frame: Baseline, rehabilitation discharge, month 3, month 6
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CO-OP | Attention Control
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline Scores | 65.27 (2.80) | 62.60 (4.28)
  Discharge Scores | 86.80 (3.27) | 80.53 (5.73)
  Month 3 | 109.69 (2.61) | 91.23 (7.48)
  Month 6 | 113.31 (2.48) | 95.27 (7.60)
Statistical Analysis 1: Comparison: CO-OP vs Attention Control; All analyses were performed using the intent-to-treat principle so that comparisons were made according to the assigned intervention group regardless of study completion; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — a priori threshold set at p<0.05; F(3,74)=4.37 P-values were calculated using mixed model analyses and controlled for stoke severity as a covariate; Cohen's d effect size at month 6 = 1.11 — Effect size was calculated using mean change scores (baseline to month 6) and standard error of change (baseline to month 6) for each group

2. Secondary Outcome: Difference in Executive Function- Inhibition, CWI (Color Word Interference Inhibition Scale)
Description: Difference mean scaled scores (Color Word Interference Inhibition Scale) between groups over time using mixed effects models.
  The Color Word Interference Inhibition Scale raw scores are converted to norm-referenced scaled scores adjusted for age and education. These scores are aligned with a population mean of 10, and standard deviation of 3. Higher scores indicate better executive function. Scaled scores were generated at baseline, month 3, and month 6 for each participant, and mean scaled scores were computed for each group at each time point.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CO-OP | Attention Control
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline Scores | 4.85 (1.14) | 4.00 (0.77)
  Month 3 Scores | 8.73 (3.00) | 4.40 (1.37)
  Month 6 Scores | 8.20 (1.13) | 3.67 (1.11)
Statistical Analysis 1: Comparison: CO-OP vs Attention Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis — a priori threshold set at p<0.05; F(2,34)=2.55; Cohen's d effect size at month 6 = .76 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Difference in Executive Function - Cognitive Flexibility, CWI (Color Word Interference Switching Scale)
Description: Difference between groups in mean scaled scores (Color Word Interference Switching Scale) over time using mixed effects models.
  The Cognitive Flexibility Scale raw scores were converted to norm-referenced scaled scores adjusted for age and education. These scores are aligned with a population mean of 10, and standard deviation of 3. Higher scores indicate better executive function. Scaled scores were generated at baseline, month 3, and month 6 for each participant, and mean scaled scores were computed for each group at each time point.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CO-OP | Attention Control
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline Scores | 3.69 (0.65) | 2.73 (0.61)
  Month 3 Scores | 8.82 (0.81) | 3.00 (0.93)
  Month 6 Scores | 8.20 (0.73) | 2.78 (0.93)
Statistical Analysis 1: Comparison: CO-OP vs Attention Control; All analyses were performed using the intent-to-treat principle so that comparisons were made according to assigned intervention group regardless of study completion; Test type: Superiority or Other; p = .002, Mixed Models Analysis — a priori threshold set at p<0.05; F(2,34)=7.83; Cohen's d effect size at month 6 = 1.23 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Differences in Apathy Symptoms Between Groups Over Time
Description: Difference in mean Apathy Evaluation Scale total scores were examined between groups over time using repeated measures fixed effects models.
  The Apathy Evaluation Scale measures lack of motivation or interest in goal-directed activities. The scale has 18 items yielding a total score of 18 (indicating absence of apathy) to 72 (indicating severe apathy). Total scores were generated for each participant at each time, and mean scores were computed for each group at each time point.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CO-OP | Attention Control
Number analyzed (Participants) | 15 | 15
units on a scale
  Baseline Scores | 25.79 (2.04) | 25.18 (1.32)
  Month 3 Scores | 25.18 (1.65) | 34.13 (4.70)
  Month 6 Scores | 21.38 (1.34) | 29.00 (4.82)
Statistical Analysis 1: Comparison: CO-OP vs Attention Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .04, repeated measures fixed effects model — a priori threshold set at <0.05; F(2,28)=3.61; Cohen's d effect size at month 6 = 0.70 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | CO-OP | Attention Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes